CLINICAL TRIAL: NCT04203368
Title: Efficacy of Adenosine Versus Verapamil for Management of Supraventricular Tachycardia Post- Coronary Artery Bypass Grafting: a Randomized Double Blinded Trial
Brief Title: Adenosine Versus Verapamil for Management of Supraventricular Tachycardia Post- Coronary Artery Bypass Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Assistant professor of Anaesthesiology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 62/ 2019
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Supraventricular Tachycardia
Keywords: SVT; CABG; verapamil; adenosine
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Adenosine; Verapamil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adenosine group (Active Comparator): patients received IV adenosine 6 mg bolus then wait 2 minutes, if it failed to return to sinus rhythm then another 12 mg IV bolus of adenosine was administered, if supraventricular tachycardia persisted then the patient was shifted to verapamil
  Interventions: Drug: adenosine
- verapamil group (Sham Comparator): patients received IV verapamil 5mg bolus slowly over 2 minutes followed by a second IV bolus dose of 5 mg ,10 minutes after the initial dose in case of persistence of supraventricular tachycardia (SVT). If SVT persisted, the patient was shifted to adenosine
  Interventions: Drug: verapamil

INTERVENTIONS:
Drug: adenosine — patients received IV adenosine 6 mg bolus then wait 2 minutes, if it failed to return to sinus rhythm then another 12 mg IV bolus of adenosine was administered, if supraventricular tachycardia persisted then the patient was shifted to verapamil.
  Arms: adenosine group
Drug: verapamil — patients received IV verapamil 5mg bolus slowly over 2 minutes followed by a second IV bolus dose of 5 mg ,10 minutes after the initial dose in case of persistence of supraventricular tachycardia (SVT). If SVT persisted, the patient was shifted to adenosine
  Arms: verapamil group

SUMMARY:
This prospective study was conducted in 268 patients aged from 65-70 years posted for coronary artery bypass grafting. Patients were randomly allocated to either adenosine or verapamil(control) groups. In the adenosine group, patients received IV adenosine 6 mg bolus then wait 2 minutes, if it failed to return to sinus rhythm then another 12 mg IV bolus of adenosine was administered, if supraventricular tachycardia persisted then the patient was shifted to verapamil. In verapamil group, patients received IV verapamil 5mg bolus slowly over 2 minutes followed by a second IV bolus dose of 5 mg ,10 minutes after the initial dose in case of persistence of supraventricular tachycardia (SVT). If SVT persisted, the patient was shifted to adenosine. The efficacy of the study drug, ICU stay length, systolic blood pressure, hospital- stay length, duration of extubation, the total dose of the study drug used, the total cost of the study drugs and the incidence of adverse events were recorded.

DETAILED DESCRIPTION:
Written informed consent was obtained from every patient. This prospective, double-blind, parallel-group clinical trial was conducted in 268 patients. The following inclusion criteria were used: (1) RCT; (2) adult (age: 65-70 years) patients with ASA physical status II and III, scheduled for elective isolated CABG; (3) use of adenosine versus verapamil for treatment of postoperative supraventricular tachycardia; (4) the efficacy was a mandatory outcome measurement ; (5) Ejection fraction 50-60%; (6) Absence of any associated comorbidities or history of myocardial infarction. Patient with impaired cerebral Perfusion, hemodynamic instability arrhythmias other than PSVT were excluded.

Anesthesia management was standardized to minimize any effect of anesthetic type on hemodynamics. Premedication with midazolam was limited to a maximum of 0.05 mg/kg. Anesthesia was induced with 12 μg/kg fentanyl, 5-7 mg/kg thiopental sodium, and 0.15 mg/kg pancuronium and was maintained with 1-2.0% isoflurane. Heart rate and blood pressure were maintained within 20% of the baseline values. Anticoagulation was achieved with heparin 300 U/kg administered into the right atrium to maintain an activated clotting time above 480 s. Cardiopulmonary bypass (CPB) was conducted with non-occlusive roller pumps, membrane oxygenators, arterial line filtration, and cold blood-enriched hyperkalemic arrest. The CPB circuit was primed with 1.8 l lactated Ringer's solution and 50 ml of 20% mannitol. Management of CPB included systemic hypothermia (to an esophageal temperature of 32°C) during aortic cross-clamping, targeted mean perfusion pressure between 60 and 80 mmHg, and pump flow rates of 2.2 l/min/m2. Myocardial protection was achieved with antegrade cold blood cardioplegia. A 32-μm filter (Avecor Affinity, Minneapolis, MN, USA) was used in the arterial perfusion line. Before separation from CPB, patients were warmed to 36-37°C. After separation from CPB, heparin was neutralized with protamine sulfate and 1 mg/100 U heparin to reach an activated clotting time within 10% of baseline. All patients were transferred to the ICU after surgery.

Patients were randomly allocated to either adenosine or verapamil(control) groups according to a computer-generated randomization code, with allocation ratio 1:1. Opaque sealed envelopes were prepared according to the randomization schedule, and were opened by a clinician not involved in any part of the study. Upon arrival at the ICU, a standardized protocol for postoperative care was implemented for all patients by well-trained nurses supervised 1:1and by the ICU consultants. The study medications were calculated and prepared by ICU nurses who were not a part of the research team. Both end-point assessors of the outcomes and patients were blinded to the study drugs. All staff were blinded to treatment allocation excluding the ICU consultant and resident who were not part of the research team.

To ensure blinding of study drug administration, the medication vials were kept in opaque bags. Trial bags were blinded and marked with a unique number. The allocation of trial drugs was determined by the web-based randomization system by the allocation of the bag number.

In the adenosine group, patients received IV adenosine 6 mg bolus then wait 2 minutes, if it failed to return to sinus rhythm then another 12 mg IV bolus of adenosine was administered, if supraventricular tachycardia persisted then the patient was shifted to verapamil. In verapamil group, patients received IV verapamil 5mg bolus slowly over 2 minutes followed by a second IV bolus dose of 5 mg ,10 minutes after the initial dose in case of persistence of supraventricular tachycardia (SVT). If SVT persisted, the patient was shifted to adenosine.

All patients were routinely extubated when deemed clinically appropriate according to the local ICU protocol, by ICU staff, when the patient was able to maintain spontaneous breathing for 48 h, according to normal weaning parameters, after which they were encouraged to sit on a chair and mobilize with the assistance of health care providers in the ICU then the physiotherapist became responsible for improving mobility and rehabilitation of the patients till discharge from the hospital. Systolic blood pressure and heart rate were continuously monitored during drug administration and 30 minutes after conversion to sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

* RCT
* 65-70 years old
* elective CABG

Exclusion Criteria:

* impaired cerebral Perfusion
* hemodynamic instability
* arrhythmias other than PSVT

Ages: 65 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-11-22 (Actual)

PRIMARY OUTCOMES:
efficacy of the study drug | 5 days postoperative
  cardioversion to sinus rhythm

SECONDARY OUTCOMES:
ICU stay | 2 days postoperative
  ICU stay duration
duration of extubation | 6-12 hours postoperative
  extubation time

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt